CLINICAL TRIAL: NCT05602480
Title: Phase I Clinical Trial to Evaluate the Safety and Explore the Immunogenicity of a Candidate PCV13 in Healthy People Aged 2 Months (Minimum 6 Weeks) and Above
Brief Title: Phase I Clinical Trial of a Candidate PCV13 in Healthy People
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan BravoVax Co., Ltd. (Industry)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other); Liaoning Chengda Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLI-09-I-2020001
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Pneumococcal Infections
Keywords: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One arm, open label in subjects aged 3 months and above; Randomized, blinded and active comparator in subjects aged 2 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 1A (Experimental): Subjects received one dose of PCV13 at 18 years of age and above.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 2A (Experimental): Subjects received one dose of PCV13 at 6~17 years of age.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 3A (Experimental): Subjects received one dose of PCV13 at 2~5 years of age.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 4A (Experimental): Subjects received two doses of PCV13 at 12~23 months of age.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 5A (Experimental): Subjects received three doses of PCV13 at 7~11 months of age.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 6A (Experimental): Subjects received four doses of PCV13 at 3 months of age.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 6B (Experimental): Subjects received four doses of PCV13 at 2 months of age (At least 6 weeks old).
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 6C (Active Comparator): Subjects received four doses of control PCV13 at 2 months of age (At least 6 weeks old).
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 7A (Experimental): Subjects received four doses of PCV13 at 2 months of age (At least 6 weeks old).
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 7B (Active Comparator): Subjects received four doses of control PCV13 at 2 months of age (At least 6 weeks old).
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine — 0.5mL, Intramuscular
  Other Names: PCV13
  Arms: 1A; 2A; 3A; 4A; 5A; 6A; 6B; 7A
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine — 0.5mL, Intramuscular
  Other Names: Prevnar 13
  Arms: 6C; 7B

SUMMARY:
Streptococcus pneumoniae is a major cause of morbidity and mortality in children worldwide, resulting in up to 1 million pediatric deaths every year. Since the licensure of PCV7, PCV10, PCV13 and PCV15, the reported overall decline in invasive pneumococcal disease in hospitalized children younger than 5 years is approximately 60% around the world.

This is a single center, blinded, randomized, positive-controlled phase I clinical trial to evaluate the safety and explore the immunogenicity of a candidate PCV13 in healthy people aged 2 months (minimum 6 weeks) and above.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy the age requirements of the clinical trial; willing to provide proof of identity;
* Subjects or guardians must provide informed consent forms with personal signature and date;
* Male and female of childbearing age should agree to take effective contraception measures;
* Subjects or guardians can obey the requirements of the clinical study;
* Axillary temperature below 37.3 °C.

Exclusion Criteria:

* Laboratory indicators (expect those have no clinical significance) out of normal ranges required;
* Received any pneumococcal vaccine;
* Allergic history to any drugs, vaccine or vaccine-related component;
* Infants with congenital malformations, developmental disorders, genetic defects, or severe malnutrition;
* Infants diagnosed with pathological jaundice that lasts for 2~4 weeks and occurs repeatedly;
* Breast-feeding or pregnant women, or positive U-HCG;
* High blood pressure uncontrolled by medication;
* Known or suspected immune deficiency or immune suppression;
* Serious congenital malformation, history of organ resection or serious chronic illness;
* Received blood products or intravenous immunoglobulin (except Hepatitis B immunoglobulin);
* History of clinic-proven or serology-proven infectious disease especially caused by streptococcus pneumoniae;
* History of convulsions, epilepsy or encephalopathy or a family history of mental illness;
* A vaccination-related contraindications that other investigator believes;
* Plans to participate in or is participating in any other clinical study;
* Any other factors judged by investigator that may interfere subject's compliance with the protocol.

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of adverse reactions | within 30 minutes post each vaccination
  Occurrence of AEs on vaccination site (local) and non-vaccination site (systemic) of each subject
Safety in terms of adverse events | within 7 days post each vaccination
  Occurrence of solicited AEs of each subject
Safety in terms of adverse events | within 30 days post each vaccination
  Occurrence of non-solicited AEs of each subject
Safety in terms of SAEs | within 6 months post last vaccination
  Occurrence of SAEs of each subject
Safety in terms of laboratory-based AEs | within 4 days post each vaccination
  Occurrence of laboratory-based AEs in subjects of 2 years old and above(Arm 1A-3A)

SECONDARY OUTCOMES:
Immunogencity in terms of seropositivity rates by ELISA | 30 days post basic vaccination
  Seropositivity rates of serotype-specific pneumococcal IgG antibody in subjects of each age group
Immunogencity in terms of GMC by ELISA | 30 days post basic vaccination
  GMC of serotype-specific pneumococcal IgG antibody in subjects of each age group
Immunogencity in terms of subjects with IgG concentrations ≥1.0 µg/mL | 30 days post basic vaccination
  Percentage of subjects with serotype-specific IgG concentrations ≥1.0 µg/mL
Immunogencity Comparison with control vaccine group | 30 days post basic vaccination
  Comparison of the seropositivity rates, GMC of serotype-specific pneumococcal IgG antibody and the Percentage of subjects with serotype-specific IgG concentrations ≥1.0 µg/mL in subjects aged 2 months of Experimental group and Control group

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangtan Maternal and Child Health Hospital, Xiangtan, Hunan, China